CLINICAL TRIAL: NCT01577069
Title: Predictive Factors of the Treatment Failure in HCV Mono-infected Patients Treated With Pegylated-interferon/Ribavirin/Telaprevir.
Brief Title: Predictive Factors of the Treatment Failure in Hepatitis C Virus (HCV) Infected Patients Treated With Telaprevir
Acronym: GENUPI
Status: Completed | Type: Observational
Sponsor: Association HGE CHU Bordeaux Sud (Other)
Collaborators: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: UDPS-100211
Record Dates: First submitted 2012-04-12; First posted 2012-04-13 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C; Direct Antiviral agent (DAA); Ultra-deep pyrosequencing; Single polynucleotide polymorphisms; Treatment-resistant mutants; Hepatitis C Virus Protease Inhibitor
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to

1- detect and quantify HCV-PI resistant mutants with ultra-deep pyrosequencing (UDPS) technology, 2 - detect SNPs in P-glyocoprotein and CYP3A genes, in HCV mono-infected patients under/after Telaprevir treatment.

ELIGIBILITY:
Inclusion Criteria:

* HCV mono-infected subjects
* Age > 18 years

Exclusion Criteria:

* HBV co-infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCV mono-infected patients treated in the Hepatology Unit of Pr Victor de Lédinghen (Hôpital du Haut-Lévêque, Pessac)
Sampling Method: Non-Probability Sample
Enrollment: 73 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
virological resitance | 12 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Victor de lédinghen, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Hôpital du haut-Lévêque, Pessac, France